CLINICAL TRIAL: NCT05623293
Title: Prognostic Predictors of Cardiovascular and Ophthalmologic Outcomes in Patients With Carotid Artery Stenosis Undergoing Carotid Endarterectomy With Regional Anesthesia - A Prospective Study
Brief Title: Ophthalmologic Outcomes in Patients With Carotid Artery Stenosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidade do Porto (Other)
Collaborators: Hospital Sao Joao (Other)
Responsible Party: Principal Investigator, João Rocha Neves, Principal Investigator, Universidade do Porto
Other Study IDs: 163-21
Record Dates: First submitted 2021-08-15; First posted 2022-11-21 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Choroid Disease; Carotid Stenosis; Carotid Atherosclerosis; Retinal Disease
Keywords: Carotid endarterectomy; Optimal coherence tomography,
MeSH Terms: conditions — Choroid Diseases; Carotid Stenosis; Carotid Artery Diseases; Retinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Carotid endarterectomy: he population corresponds to patients submitted to elective CEA. Consecutive patients from a tertiary referral center who undergo CEA for carotid artery stenosis (CS) under regional anesthesia will be prospectively recruited from September 2021 - December 2022. The expected patient follow-up will be of 2years.
  Interventions: Diagnostic Test: eye - Optcial coherence tomography

INTERVENTIONS:
Diagnostic Test: eye - Optcial coherence tomography — pre and postoperative

SUMMARY:
The retinal vessels have been shown to reflect vascular changes inherent to systemic pathologies, even when no ocular disease is identified. As such, the eye's vasculature is ableto serve as a window to the vascular health of the human body and a means of assessing systemic endothelial function. Optical coherence tomography angiography (OCTA) employs optical means to image all the retinal vascular layers and the choroid, providing an extremely detailed image of the microvascular network in a fast, reproducible and totally non-invasive way. As such, it is currently the best non-invasive way of having an image of human capillaries. Recently, OCTA has been used to study the retinal vessels' structure and function in several cardiovascular diseases. As an example of its predictive potential, reduced retinal microvascular density has been associated with the cardiovascular risk profile in patients admitted to the hospital for an acute coronary syndrome. Recent studies have also shown the retinal microvasculature density to be reduced in patients with carotid artery disease (CAD), namely carotid stenosis, and that endarterectomy increases retinal flow and vessel density.

DETAILED DESCRIPTION:
The authors hypothesize that FGF-23, GDF-15, VEGF-A, MMP-9 and retinal/choroidal microvascular density could predict cerebral ischemia, postoperative complications, long term major cardiovascular events and short term ophthalmologic alterations particularly in patients developing symptomatic neurologic ischemia after circulation shutdown.

The purpose of this study is to compare different cardiac risk scores in carotid endarterectomy. The main aim of this study is to test the risk factors individually and determine its discriminatory ability. Combinations of traditional preoperative risk factors and scores will be evaluated to enhance the assessment of major adverse cardiac events in vascular surgery patients.

Establish and validate biomarkers that improve the predictive value of current risk stratification models for patients benefiting from carotid revascularization, outperform existing biomarkers, and reach clinical application standards.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive carotid stenosis

Exclusion Criteria:

* blind patients
* Radic stenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is a non-interventional prospective cohort study. The population corresponds to patients submitted to elective CEA. Consecutive patients from a tertiary referral center who undergo CEA for carotid artery stenosis (CS) under regional anesthesia will be prospectively recruited from September 2021 - December 2022. The expected patient follow-up will be of w year
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Stroke | 30 days
  diagnosed by Computer tomography and clinical examation
optical coherence tomography - Angio | 15 days before surgery
  Vessel density and distribution
optical coherence tomography - Angio | 24h after surgery
  Vessel density and distribution
optical coherence tomography - Angio | 30 days after surgery
  Vessel density and distribution
optical coherence tomography - Angio | one year after surgery
  Vessel density and distribution

SECONDARY OUTCOMES:
Restenosis | 2 months
  ultrasound defined - internacal carotid Velocity superior to 180 cm/s; or 250 cm/s

CONTACTS AND LOCATIONS:
Locations (1):
- Joao Rocha-Neves, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No
Publications

REFERENCES:
- [Background] Nakazawa T. Ocular Blood Flow and Influencing Factors for Glaucoma. Asia Pac J Ophthalmol (Phila). 2016 Jan-Feb;5(1):38-44. doi: 10.1097/APO.0000000000000183. PMID 26886118